CLINICAL TRIAL: NCT05051176
Title: Prevalence of Diastasis m. Rectus Abdominis and Pelvic Floor Muscle Dysfunction in Postpartum Women
Brief Title: Prevalence of Diastasis m. Rectus Abdominis in Postpartum Women
Status: Completed | Type: Observational
Sponsor: Pavol Jozef Safarik University (Other)
Responsible Party: Principal Investigator, Rastislav Dudič, MD, PhD., Faculty of Medicine, Pavol Jozef Safarik University
Other Study IDs: 4168/2021/ODDZ-11065
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Diastasis of m. Rectus Abdominis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2D usg and 3D/4D usg — IRD distance measured by a linear probe 2D usg. Pelvic floor muscle morphometry measured by 3D/4D usg

SUMMARY:
This study will evaluate the prevalence of diastasis m. rectus abdominis after delivery.

Relationship of Diastasis Recti Abdominis with urine leakage, pelvic floor muscle function and morphometry in postpartum women.

DETAILED DESCRIPTION:
Evaluation of the width of the linea alba within the evaluation of diastasis of the rectus abdominis by 2D USG relation to pelvic floor muscle function (strength and endurance of pelvic floor muscles) and pelvic floor muscle morphometry by 3D/4D USG .

ELIGIBILITY:
Inclusion Criteria:

* Women from six weeks to up to 6 months after birth, age over 18 years old.

Exclusion Criteria:

* Psychiatric illness, postpartum depression, non-cooperation. Neurological diseases conditions after a stroke, a history of brain injury, significant visual and hearing damage, confirmed by neurological examination. Serious internal, orthopedic and oncological diseases. Disagreement with inclusion in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from six weeks to up to 6 months after birth, age over 18 years old.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of Diastasis Recti Abdominis in Postpartum Women. | Six weeks to up to 6 months after birth
  IRD distance measured by a linear probe 2D usg, 4.5 cm above the navel, 4.5 cm below the navel. At rest, and when raising the lower limbs.

SECONDARY OUTCOMES:
Relationship of Diastasis Recti Abdominis with urine leakage, pelvic floor muscle function and morphometry in postpartum women. | Six weeks to up to 6 months after birth.
  Occurrence of stress urinary incontinence using the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-UI SF).
Relationship between Diastasis Recti Abdominis and back pain in postpartum women. | Six weeks to up to 6 months after birth.
  Occurrence of low back pain using the Oswestry Disability Index (ODI).

CONTACTS AND LOCATIONS:
Overall Officials: Rastislav Dudič, PhD, Principal Investigator — Department of Gynecology and Obstetrics, Medical Faculty, PJ Safarik University, Kosice, Slovakia; Magdalena Hagovska, Prof,PhD, Study Director — KFBLR, Medical Faculty, PJ Safarik University, Kosice, Slovakia; Jan Svihra, Prof,MD,PhD., Study Director — Department of Urology, Institution, Comenius University Bratislava, Slovakia
Locations (1):
- PJ Safarik University, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No